CLINICAL TRIAL: NCT04624438
Title: Central and Peripheral Changes in Quadriceps Femoris Function After Different Types of Isometric Strength Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Collaborators: University of Primorska, Faculty of Health Sciences (Unknown)
Responsible Party: Principal Investigator, Dragan Mirkov, Professor Dr., University of Belgrade
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 02-672-2/09-04-2015
Record Dates: First submitted 2020-11-02; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Quadriceps Muscle Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Electromyostimulation - EMS (Experimental): Experimental group comprised of healthy young adults that undergoes unilateral isometric training using electromyostimulation over quadriceps femoris
  Interventions: Other: Isometric training with electromyostimulation
- Voluntary activation - VOLUNTARY (Experimental): Experimental group comprised of healthy young adults that undergoes unilateral isometric training based on voluntary activation of quadriceps femoris
  Interventions: Other: Isometric training with voluntary activation
- Combination of EMS and VOLUNTARY - COMBINED (Experimental): Experimental group comprised of healthy young adults that undergoes unilateral isometric training that combines electromyostimulation and voluntary activation of quadriceps femoris.
  Interventions: Other: Isometric training with combination of electromyostimulation and voluntary activation
- Control group - CONTROL (No Intervention): Group of healthy young adults who received no intervention.

INTERVENTIONS:
Other: Isometric training with electromyostimulation — Each training session (18 in total) consisted of forty 4-s contractions separated by 20 s inter-contraction intervals. The exercise intensity was close-to-identical among the sessions (60 %MVC). The force intensity was determined individually during pretest where EMS was delivered at maximal tolerable dose. Electrical stimulation was 6.25-second long and was followed by a rest period of 20-second (duty cycle 15%). Stimulation characteristics were selected among the "Compex" commercially available strength programs. The stimulation intensity was monitored on-line and determined by the subject at the start of each EMS session according to his/her pain threshold to produce a force corresponding to at least 60% of the pretest MVC score.
  Arms: Electromyostimulation - EMS
Other: Isometric training with voluntary activation — Each training session (18 in total) consisted of forty 4-s contractions separated by 20 s inter-contraction intervals. The exercise intensity was close-to-identical among the sessions (60 %MVC). Participants were required to reach the proscribed force level only through voluntary activation of QF. To attain the same contraction/rest ratio as in EMS, automated audible signals were delivered in accordance with the contraction-rest pattern produced by the muscle stimulation device. To ensure participants produced 60% of individual MVC during each contraction the force level was measured with a force transducer and real-time feedback was provided on a computer screen.
  Arms: Voluntary activation - VOLUNTARY
Other: Isometric training with combination of electromyostimulation and voluntary activation — Each training session (18 in total) consisted of forty 4-s contractions separated by 20 s inter-contraction intervals. The exercise intensity was close-to-identical among the sessions (60 %MVC). The proscribed force level was reached by the simultaneous action of EMS and VOLUNTARY. Each contraction was 6.25-second long and was followed by a rest period of 20-second (duty cycle 15%). Electrical stimulation corresponded to 30% of MVC, while the remaining 30% was achieved through voluntary muscle activation. To ensure participants produced a force corresponding to 60% of MVC during each contraction the force level was measured with a force transducer and real-time feedback was provided on a computer screen.
  Arms: Combination of EMS and VOLUNTARY - COMBINED

SUMMARY:
The purpose of this investigation is to examine the effects of 6-week unilateral isometric training interventions over quadriceps femoris on maximal strength and RFD-SF parameters and cortical excitability. Isometric strength training involved either electromyostimulation, voluntary activation, or the combination of both. The second aim is to investigate the potential cross-over effect on a non-trained leg.

DETAILED DESCRIPTION:
A longitudinal pre-post design with random assignment of the participants to one of three experimental groups or the control group was used. Quadriceps femoris (QF) function and cortical excitability were assessed on four occasions: prior to the intervention (pre-test), after 3 weeks of training (served for the adjustment of exercise intensity), after 6 weeks of training (post-test), and three weeks after the competition of training intervention (detraining) (Figure 1). Isometric strength training involves activation of QF applying EMS, VOLUNTARY, or the combination of both EMS and VOLUNTARY (COMBINED). The pre-test also served to familiarize participants with the training protocols and to determine the intensity of EMS needed to achieve 60%MVC. Quadriceps femoris (QF) function was assessed by MVC and RFD-SF. Cortical excitability was assessed with transcranial magnetic stimulation applied over the M1 region. Prior to the pretest, body mass and percent of body fat were assessed using a bioelectric impedance method (In Body 720; USA) and body height with a standard stadiometer. After the pretest, the participants were randomly assigned to either one of the experimental groups (EMS, VOLUNTARY, or COMBINED) and the control group (CONTROL). Experimental groups performed unilateral isometric strength training three times per week for 6 weeks. All participants were advised to refrain from all resistance training targeting the legs between pre-test and post-test.

ELIGIBILITY:
Inclusion Criteria:

* young healthy, physically active participants of both genders

Exclusion Criteria:

* no history of injuries, muscle-skeletal or neurological disease, or medications intake

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
MVC | Baseline
  Maximal isometric force and Rate of Force Development of quadriceps femoris muscle during isometric contractions with maximal effort
MVC | After 3 weeks
  Maximal isometric force and Rate of Force Development of quadriceps femoris muscle during isometric contractions with maximal effort
MVC | After 6 weeks
  Maximal isometric force and Rate of Force Development of quadriceps femoris muscle during isometric contractions with maximal effort
MVC | After 9 weeks
  Maximal isometric force and Rate of Force Development of quadriceps femoris muscle during isometric contractions with maximal effort
The slope of the rate-of-force development scaling factor (RFD-SF) | Baseline
  The slope of the relationship (RFD-SF) between muscle force and rate of force development during rapid isometric contractions of varying intensities
The slope of the rate-of-force development scaling factor (RFD-SF) | After 3 weeks
  The slope of the relationship (RFD-SF) between muscle force and rate of force development during rapid isometric contractions of varying intensities
The slope of the rate-of-force development scaling factor (RFD-SF) | After 6 weeks
  The slope of the relationship (RFD-SF) between muscle force and rate of force development during rapid isometric contractions of varying intensities
The slope of the rate-of-force development scaling factor (RFD-SF) | After 9 weeks
  The slope of the relationship (RFD-SF) between muscle force and rate of force development during rapid isometric contractions of varying intensities
Motor Evoked Potentials (MEP) | Baseline
  MEPs were elicited in quadriceps femoris by transcranial magnetic stimulation (TMS) over M1 area. Motor cortex excitability was estimated by measuring the MEP amplitude (Input-Output, IO) peak to peak, caused by 20 randomized individual TMS stimulates with 100% (IO1), 120% (IO2) and 130% (IO3) of active motor threshold (AMT) intensity.
Motor Evoked Potentials (MEP) | After 3 weeks
  MEPs were elicited in quadriceps femoris by transcranial magnetic stimulation (TMS) over M1 area. Motor cortex excitability was estimated by measuring the MEP amplitude (Input-Output, IO) peak to peak, caused by 20 randomized individual TMS stimulates with 100% (IO1), 120% (IO2) and 130% (IO3) of active motor threshold (AMT) intensity.
Motor Evoked Potentials (MEP) | After 6 weeks
  MEPs were elicited in quadriceps femoris by transcranial magnetic stimulation (TMS) over M1 area. Motor cortex excitability was estimated by measuring the MEP amplitude (Input-Output, IO) peak to peak, caused by 20 randomized individual TMS stimulates with 100% (IO1), 120% (IO2) and 130% (IO3) of active motor threshold (AMT) intensity.
Motor Evoked Potentials (MEP) | After 9 weeks
  MEPs were elicited in quadriceps femoris by transcranial magnetic stimulation (TMS) over M1 area. Motor cortex excitability was estimated by measuring the MEP amplitude (Input-Output, IO) peak to peak, caused by 20 randomized individual TMS stimulates with 100% (IO1), 120% (IO2) and 130% (IO3) of active motor threshold (AMT) intensity.

SECONDARY OUTCOMES:
The linearity of the rate-of-force development scaling factor (RFD-SF) relationship | Baseline
  The linearity, described by coefficient of determination (r-squared) of the relationship (RFD-SF) between muscle force and rate of force
The linearity of the rate-of-force development scaling factor (RFD-SF) relationship | After 3 weeks
  The linearity, described by coefficient of determination (r-squared) of the relationship (RFD-SF) between muscle force and rate of force
The linearity of the rate-of-force development scaling factor (RFD-SF) relationship | After 6 weeks
  The linearity, described by coefficient of determination (r-squared) of the relationship (RFD-SF) between muscle force and rate of force
The linearity of the rate-of-force development scaling factor (RFD-SF) relationship | After 9 weeks
  The linearity, described by coefficient of determination (r-squared) of the relationship (RFD-SF) between muscle force and rate of force
M-wave | Baseline
  The tracing of the earliest electromyography (EMG) response to the stimulation of femoral nerve
M-wave | After 3 weeks
  The tracing of the earliest electromyography (EMG) response to the stimulation of femoral nerve
M-wave | After 6 weeks
  The tracing of the earliest electromyography (EMG) response to the stimulation of femoral nerve
M-wave | After 9 weeks
  The tracing of the earliest electromyography (EMG) response to the stimulation of femoral nerve

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sport and Physical Education, University of Belgrade, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Data will be available after a request to PI
Supporting Information: Study Protocol, SAP
Time Frame: Six months after the completion of the study
Access Criteria: No specific sharing access criteria